CLINICAL TRIAL: NCT03729323
Title: Nursing Consultation Based on Motivational Interviewing as a Strategy for the Control of Type 2 Diabetes Mellitus and Systemic Arterial Hypertension in Primary Healthcare: A RANDOMIZED CLINICAL TRIAL
Brief Title: Motivational Interviewing in the Control of Arterial Hypertension and Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Nossa Senhora da Conceicao (Other)
Responsible Party: Principal Investigator, Daniel Demétrio Faustino da Silva, Dokter Odontologist, Hospital Nossa Senhora da Conceicao
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Grupo Hospitalar Conceicao
Record Dates: First submitted 2018-10-07; First posted 2018-11-02 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Type 2 Diabetes Mellitus; Systemic Arterial Hypertension
Keywords: Motivational Interviewing; Type 2 Diabetes Mellitus; Systemic Arterial Hypertension; Chronic Diseases; Self-care
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Chronic Disease | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Clinical-behavioral
Who Masked: Participant, Outcomes Assessor
Masking Description: Double Blind. The person responsible for randomizing and allocating research subjects, outcome assessors and those responsible for data analysis will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Motivational Interviewing (Experimental): INTERVENTION GROUP: In this group, Diabetics and Hypertensives will attend two Nursing Consultation sessions based on the assumptions and techniques of Motivational Interviewing with a certified nurse with specific 20-hour theoretical and practical training for this approach style.
  Interventions: Behavioral: Motivational interviewing
- Nursing Consultation (Active Comparator): CONTROL GROUP: In this group, Diabetics and Hypertensives will attend two conventional nursing consultation sessions aimed at self-care, with a untrained nurse for the use of motivational interviewing, based on the recommendations of the Primary Care Strategy Notebooks for the care of chronic conditions in Diabetes Mellitus and Arterial Hypertension and the SSC-GHC Institutional Protocol for SAH and DM2 Patient Care.
  Interventions: Behavioral: Nursing Consultation

INTERVENTIONS:
Behavioral: Motivational interviewing — In Diabetes and hypertension, nursing consultations to support the care should be focused on their educational component the orientation of measures that prove to reduce blood pressure, improve the glycemic indices, the lipid profile and the Cardiovascular risk classification, among them: adherence to drug therapy, proper diet, body weight maintenance, stimulating active life and regular physical exercise, reducing alcoholic beverage consumption, reducing stress and abandoning Smoking. In this group, these care will be addressed based on the principles and techniques of the Motivational Interviewing.
  Arms: Experimental: Motivational Interviewing
Behavioral: Nursing Consultation — In Diabetes and hypertension, nursing consultations to support the care should be focused on their educational component the orientation of measures that prove to reduce blood pressure, improve the glycemic indices, the lipid profile and the Cardiovascular risk classification, among them: adherence to drug therapy, proper diet, body weight maintenance, stimulating active life and regular physical exercise, reducing alcoholic beverage consumption, reducing stress and abandoning Smoking. In this group, these care will be approached in a conventional manner, as routine of the services, based on the recommendations of the Primary Care Strategy Notebooks for the care of chronic conditions in DM2 and SAH and the SSC-GHC Institutional Protocol for SAH and DM2 Patient Care.
  Arms: Nursing Consultation

SUMMARY:
The goal of this study is to evaluate the effectiveness of Nursing Consultation based on the assumptions and techniques of Motivational Interviewing for the control of Type 2 diabetes mellitus with associated diagnosis of Systemic Arterial Hypertension in primary healthcare.

DETAILED DESCRIPTION:
Type 2 Diabetes Mellitus and Systemic Arterial Hypertension are major challenges to health systems worldwide, and control, adherence and promotion of self-care are the cornerstone of their management. In this context, an adequate therapist-patient relationship is the key to the success of these interventions in healthcare, and nurses have a recognized and outstanding role in improving adherence and care results in chronic diseases. Motivational Interviewing (MI) emerges as a skillful method of counseling that has proven to be effective in promoting changes in a wide variety of health-related behaviors, including hypertension and diabetes. Despite the increasing number of international studies in different health fields, the scientific production that assess the applicability of Motivational Interviewing to chronic diseases in the Brazilian setting is still modest. Recent studies suggest the need for further research involving the discussion and improvement of studies utilizing Motivational Interviewing in Brazil, as well as in other countries around the world, for better outlook on this area of investigation. Therefore, this study intends to contribute to this perspective and aims to investigate the effectiveness of this care strategy in individual Nursing consultations for people with DM2 and SAH who are being treated in three Primary Healthcare Clinics in the Northern Area of Porto Alegre - RS , Brazil, which are an integral part of the Grupo Hospitalar Conceição (GHC) Community Health Service (SSC). GHC treats patients from the Brazilian public health system exclusively, with universal and free access, and the SSC is comprised of 16 primary care and mental health services, caring for a population of 105,000 inhabitants in the northern and eastern areas of Porto Alegre, RS, Brazil. This will be a randomized, controlled, parallel and double-blind clinical trial to be conducted in the period from June to September, 2018.

MAIN GOAL: To evaluate the effectiveness of Nursing Consultation based on the assumptions and techniques of Motivational Interviewing in the control of Type 2 Diabetes Mellitus with associated diagnosis of Systemic Arterial Hypertension in primary healthcare.

SPECIFIC GOALS:

* To characterize participants in terms of sociodemographic and economic profile, health history, and life habits;
* To monitor and assess glycemic and pressure goals before and after intervention;
* To estimate the prevalence of adherence to drug therapy and healthy life habits among participants before and after intervention;
* To assess self-efficacy for participants' self-care before and after intervention.
* To evaluate the Level of Importance and Confidence to change unhealthy behaviors among participants with DM2 and SAH, before and after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years old or older;
* Having diagnosis of Type 2 Diabetes Mellitus and Systemic Arterial Hypertension.
* Being registered in the programmatic action of the clinics under study under risk stratum 3;

Exclusion Criteria:

* Being assessed at a risk stratum other than 3 at the time of the first meeting with the control and intervention group;
* Showing a cognitive deficit or associated diseases compromising the patient's mental faculties

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2021-03-12 (Actual)

PRIMARY OUTCOMES:
Glycated hemoglobin | 3 months after the end of two Nursing Consultation sessions as a intervention
  Mean difference between laboratory examination of glycated hemoglobin at baseline and 3 months after the end of two Nursing Consultation sessions as a intervention;
Blood pressure | 3 months after the end of two Nursing Consultation sessions as a intervention
  Mean difference of systolic and diastolic blood pressure at baseline and 3 months after the end of two Nursing Consultation sessions as a intervention;

CONTACTS AND LOCATIONS:
Locations (1):
- Nossa Senhora da Conceição Hospital, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Steffen PLS, Mendonca CS, Meyer E, Faustino-Silva DD. Motivational Interviewing in the Management of Type 2 Diabetes Mellitus and Arterial Hypertension in Primary Health Care: An RCT. Am J Prev Med. 2021 May;60(5):e203-e212. doi: 10.1016/j.amepre.2020.12.015. Epub 2021 Feb 24. PMID 33637368